CLINICAL TRIAL: NCT07394153
Title: Pacritinib For The Reduction Of Bone Marrow Fibrosis In Patients With Myelofibrosis Who Have Thrombocytopenia; A Multicenter, Open-Label, Single Arm, Phase II Exploratory Study
Brief Title: Pacritinib For Bone Marrow Fibrosis In Patients With Myelofibrosis Who Have Thrombocytopenia
Acronym: PACRIMYEL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Enfermedades Mieloproliferativas Crónicas PH Negativas (Other)
Collaborators: Swedish Orphan Biovitrum (Industry); MFAR Clinical Research S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMFIN-MF-PACRI 2401; 2025-522509-39-00 (EU CTIS Number)
Record Dates: First submitted 2026-02-02; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Myelofibrosis，MF
Keywords: Myelofibrosis; JAK2 inhibitor; FTL3 inhibitor; pacritinib; low platelet count; IRAK1 inhibitor; Philadelphia Chromosome-negative Chronic Myeloproliferative Neoplasms; Bone fibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PACRIMYEL (Experimental): Pacritinib administed 200 mg twice a day (BID)
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — All patients enrolled will receive pacritinib 200 mg twice a day (BID). The maximum daily dose will be 400 mg of pacritinib. Pacritinib dose may be reduced by one level to 100 mg BID (200 mg total daily dose), or by two levels to 100 mg once daily (QD) for management of AEs. The treatment will be continued until progressive disease, unacceptable toxic effects, the patient no longer derives benefit from treatment, patients consent withdrawal or death, whichever occurs first.

SUMMARY:
We hypothesize that pacritinib leads to modification of the myelofibrosis (MF) disease phenotype, especially related to BM fibrosis and cytopenias; due potentially to its dual effect as an inhibitor of the JAK and NFκB pathways, through its targets JAK2 and IRAK1 respectively, leading to a decrease of inflammatory cytokines and/or effects on stem/progenitor populations restoring hematopoiesis New evidence suggests that blocking simultaneously the JAK/STAT and NF-κB pathways might have a beneficial effect on aspects that only inhibition of the JAK pathway cannot achieve: partial recovery of BM histology and

PACRIMYEL is a multicenter, open-label, single arm, phase II, exploratory study including patients with MF and platelet count between 50 - 120 x 109/L. Clinic visits will occur on weeks 4, 8, 12, 24, 36 and 52 during the first year and every 12 weeks during the second year of the treatment, and pacritinib will be dispensed at every visit to the clinic.

Bone fibrosis will be assessed by biopsy and MRI imaging [mDixon Quant "(Philips), IDEAL IQ (General Electric) or qDixon (Siemens)] on weeks 24 and 52 after the first dose of study treatment. Splenomegaly and SVR (Splenic Volume Reduction) will be assessed by physical exam and MRI imaging on weeks 24 and 52 after the first dose of study treatment if splenomegaly at diagnosis. Same MRI to evaluate BM imaging will be used to measure spleen volume. Additionally, spleen size will be assessed by physical exam during the routine clinic visits. All patients should complete all efficacy assessments through Week 52, including patients who stop study treatment or have protocol-defined progressive disease prior to Week 24 and 52, unless the patient withdraws consent or dies. For patients who discontinue treatment before disease assessments on week 24 and week 52 for other reasons different than protocol-based progression of the disease (i.e. toxicity), and with no recent disease / fibrosis assessment (last BM biopsy > 12 weeks), disease and fibrosis assessments will be performed by the end of treatment visit. The trial includes the assessment of safety (AEs, comorbidities) throughout the study period at every visit.

Patient-reported symptoms through MPN-SAF TSS 2.0 will be collected screening, baseline (C1D1), and on Week 12, Week 24, Week 36, Week 52 and in 12-weeks intervals during the second year. Blood samples for translational research will be collected at screening and at week 24 for determination of cytokines.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written and voluntary informed consent.
2. Age ≥18 years
3. Patients with a confirmed diagnosis of myelofibrosis, either primary myelofibrosis (PMF) or post polycythemia vera (PPV-MF) or post essential thrombocythemia (PET-MF).
4. Patients with thrombocytopenia, delimited by platelets counts between 50 - 120 x 109/L.
5. Patients who require JAK-2 inhibitor therapy in the opinion of the investigator and are eligible to start treatment with pacritinib either in the first line (JAK2 inhibitor-naive) or in second line setting (after no response or loss of response or intolerance to one prior JAK2 inhibitor ).

   Note: patients should have recovered to grade ≤ 1 from any toxicity from previous treatment.
6. Have a Eastern Cooperative Oncology Group Performance Status (ECOG-PS) of 0 - 2.
7. Have a dynamic international prognostic scoring system (DIPSS) Intermediate-1, Intermediate-2, or High risk.
8. Peripheral blasts count < 5% and absolute neutrophil count (ANC) of ≥500/μL.
9. Adequate liver and renal function, defined by:

   1. liver transaminases, including alanine aminotransferase (ALT or GOT) and aspartate aminotransferase (AST or GOT) ≤ 3 x upper limit normal (ULN). AST/ALT ≤5 × ULN if transaminase elevation is related to MF.
   2. Total bilirubin and/or direct bilirubin ≤ 4 x ULN.
   3. Estimated glomerular filtration rate (eGFR) > 30 mL/min.
10. Adequate coagulation defined by prothrombin time/international normalized ratio and partial thromboplastin time ≤ 1.5 × ULN.
11. If fertile, willing to use effective birth control methods during the study and up to 30 days after the last dose of pacritinib.
12. Willing to undergo and able to tolerate frequent MRI during the study and BM biopsy
13. Able to understand and willing to complete symptom assessments.

Exclusion Criteria:

1. Life expectancy <6 months.
2. Splenic irradiation within the last 6 months.
3. Previously treated with pacritinib.
4. Concurrent enrollment in another interventional trial.
5. Treatment with an experimental therapy within 28 days prior to the first dose of study treatment.
6. Systemic treatment with a strong CYP3A4 inhibitor or inducer and the treatment cannot be either discontinued or switched to a different medication within 5 half-lifes prior to study entry.
7. Severe (Child-Pugh C) liver impairment.
8. Significant recent bleeding history defined as NCI CTCAE grade ≥2 within 3 months prior to first dose of study treatment, or with active bleeding, unless precipitated by an inciting event (e.g., surgery, trauma, or injury).
9. Conditions or medications that increase the risk of bleeding, except for aspirin (dosages of ≤100 mg per day). Patients treated with "direct-acting oral anticoagulants (DOACs), could be considered for inclusion (may be consulted with the Sponsor, GEMFIN).
10. Any history of CTCAE grade ≥2 dysrhythmias or non-dysrhythmia cardiac conditions within 6 months prior to the first dose of study treatment. Patients with non-dysrhythmia or non-QTc grade 2 cardiovascular conditions , may be considered for inclusion, if stable , asymptomatic and unlikely to affect patient safety.
11. QT corrected by the Fridericia method (QTcF) prolongation >480 ms or other factors that increase the risk for QTcF interval prolongation (e.g., heart failure, hypokalemia or history of long QT interval syndrome).
12. New York Heart Association Class II, III, or IV congestive heart failure.
13. Active or uncontrolled inflammatory or chronic functional bowel disorder such as Crohn's disease, inflammatory bowel disease, chronic diarrhea or constipation
14. Other malignancy within 3 years prior to treatment Day 1, other than curatively treated basal cell or squamous cell skin or corneal cancer; curatively treated carcinoma in situ of the cervix. The exception is if patients have been disease-free for at least 5 years, and are deemed by the investigator to be at low risk for recurrence of that malignancy.
15. Known seropositivity for human immunodeficiency virus. Known active hepatitis B, or C virus infection.
16. Women who are pregnant or lactating
17. Uncontrolled intercurrent illness, including, but not limited to, ongoing active infection, psychiatric illness, or social situation that, in the judgment of the treating physician, would limit compliance with study requirements.
18. Any active GI or metabolic condition that could interfere with absorption of oral medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Decrease in reticulin fibrosis in bone marrow (BM) | from baseline to week 52 after first dose of study treatment
  Measured in BM biopsy. Percentage of patients who experience a decrease of ≥1 grade in reticulin fibrosis from baseline to week 52. Definition of BM fibrosis grade will follow the European consensus that ranges from 0 (scattered, less fibrotic) to 3 (difuse and dense reticulin, more fibrotic). Patients will be classified as improvement (fibrosis decrease ≥1 grade), no change, or worsening (fibrosis increase > 1 grade).

SECONDARY OUTCOMES:
Improvement in BM fat fraction (FF) | from baseline to week 52 after first dose of study treatment
  measured by quantitative quantitative Dixon Quant MRI or equivalent. Changes in the bone marrow associated with MF, such as replacement of the bone marrow fat by fibrosis or elevated numbers of hematopoietic cells, reduce the abundance of fat. Here we will report the percentage of patient who had an improvement in the FF (increase from baseline at week 52).
red blood cell (RBC) transfusion independence | from baseline to week 24 and week 52 after first dose of study treatment
  Percentage of patients who achieved no need of RBC transfusions during at least 12 week.
  RBC transfusion independence will be reported in subgroup of patients with the changes in the Bone Marrow (by MRI and/or BM biopsy) over the first 24 and 52 weeks of treatment.
Improvement in hemoglobin level | from baseline to week 24 and week 52 after first dose of study treatment
  Percentage of patients who improve their hemoglobin levels without transfusion. Improvement was defined as a ≥ 1.5 g/dL increase in hemoglobin from baseline.
  Changes in hemoglobin level without transfusion will be reported in subgroup of patients with the changes in the Bone Marrow (by MRI and/or BM biopsy) over the first 24 and 52 weeks of treatment.
Improvement in platelet counts | from baseline to week 24 and week 52 after first dose of study treatment
  increase of platelet count (without transfusions) in comparison to baseline of above 75 x 109/L (if platelet count was between 50 - 75 109/L at baseline) or above 100 x 109/L (if platelet count was between 75 - 100 x 109/L at baseline). Alternatively, the proportion of patients who increase platelet counts ≥25% above baseline will be measured.
Myeloproliferative neoplasms (MPN) driver-gen Variant Allele Frequency (VAF) | Baseline and at Week 24 and Week 52 after the first dose of study treatment
  JAK2, CALR, and MPL genes are drivers of myelofibrosis. Their VAF could be quantified in peripheral blood or bone marrow and its circulating levels are usually correlated with the course of the disease. We aim to find the percentage of patients who reduced their VAF at week 24 and 52.
Cummulative dose | Throughout the study period, up to approximately 2 years
  the sum of all doses of pacritinib taken from the start of study treatment, taken into consideration interruptions and reductions.
Actual dose of pacritinib | Throughout the study period, up to approximately 2 years
  defined as the real average daily dose administered. For its calculation, the cumulative dose will be divided by the duration of the treatment, considering also the interruption periods.
Relative dose intensity of pacritinib | Throughout the study period, up to approximately 2 years
  Defined as the percentage of the planned dose that has been actually administered. Calculated dividing actual dose by planned dose per day.
Frequency of treatment-related adverse events | Throughout the study period, up to approximately 2 years
  number of patients who experience a treatment-related adverse event. Events will be classified and graded according to National Cancer Institute (NCI) Common Terminology Criteria (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Francisca Ferrer Marín, M.D.; Ph.D., Study Chair — Fundación Jimenez Díaz
Locations (13):
- Spain (13):
  - Hospital del Mar Barcelona, Barcelona, Barcelona
  - Hospital Universitario Vall d´Hebron, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Universitario de Jerez, Jerez de la Frontera, Cádiz
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid
  - Fundación Jimenez Díaz, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Clínico Universitario Valencia, Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No